CLINICAL TRIAL: NCT01616602
Title: Prone Versus Left-sided Colonoscopy in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dallas VA Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: DVAMC-10-098
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2011-12

CONDITIONS: Obese
Keywords: patients; presenting; elective; colonoscopy.
MeSH Terms: conditions — Obesity | interventions — Prone Position

ARMS (2):
- Left-sided Position (Placebo Comparator)
  Interventions: Other: Standard Position
- Prone Position (Experimental)
  Interventions: Other: Prone Position

INTERVENTIONS:
Other: Prone Position — Patients were asked to lay on their abdomen for their elective colonoscopy.
  Arms: Prone Position
Other: Standard Position — The traditional left-lateral decubitus position
  Arms: Left-sided Position

SUMMARY:
For obese patients, a randomized trial aimed at determining whether colonoscopy performance and patient comfort is improved if a patient is in the prone position (lay on their abdomen) versus the traditional left-sided position.

ELIGIBILITY:
Inclusion Criteria:

* BMI >30kg/m2
* Elective Colonoscopy

Exclusion Criteria:

* Patients with prior colonic resection, strictures, or known colonic or intra-abdominal malignancy.
* Patients who are scheduled to have monitored or general anesthesia for their procedure.
* Emergency colonoscopy
* Inadequate preparation of the colon as assessed during colonoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100

CONTACTS AND LOCATIONS:
Locations (1):
- Dallas VA Medical Center, Dallas, Texas, United States